CLINICAL TRIAL: NCT05282732
Title: Retrospective Analysis of Performance and Treatment Data Collected for Genius SleddFlux Filter, Ultraflux AV 600 S Filter & Genius 90 Concentrates in Acute Haemodialysis, Haemodynamically Instable Patients and Chronic Haemodialysis Patients
Brief Title: Retrospective Analysis of Performance and Treatment Data Collected for Genius SleddFlux Filter, Ultraflux AV 600 S Filter & Genius 90 Concentrates in Haemodialysis Patients
Acronym: Genius
Status: Recruiting | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: Genius-AKI-01-D
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Renal Failure; End Stage Renal Disease; Acute Renal Failure
Keywords: Hemodialysis; Genius system; Slow extended daily dialysis
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aHD: Acute haemodialysis patients
- cHD: Chronic haemodialysis patients

SUMMARY:
Retrospective analysis of performance and treatment data collected for Genius SleddFlux Filter, Ultraflux AV 600 S Filter & Genius 90 Concentrates in acute haemodialysis, haemodynamically instable patients and chronic haemodialysis patients

* to analyse performance and treatment data from patients treated with the investigational device
* to evaluate the filter characteristics for aHD (Acute haemodialysis) patients
* to evaluate the improvement of kidney function for aHD patients

ELIGIBILITY:
Inclusion Criteria:

* All patients with an indication for the extracorporeal blood treatment suffering from renal insufficiency who received all treatments, between January 2019 and December 2019, with the investigational devices have to be included in the study in chronological order.
* For aHD patients: availability of at least 3 of the 5 primary variables (daily urea, creatinine, potassium, ultrafiltration and effluent volume) for 50 % of the documented treatments.
* For cHD patients: availability of the ultrafiltration values for all treatments and at least one value for urea and creatinine per week

Exclusion Criteria:

* Simultaneous use of another filter/adsorber for another form of therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Haemodynamically instable patients in acute haemodialysis and chronic haemodialysis patients treatment with the Genius system
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Daily values for urea, Unit: mg/dl or mmol/L | During the intervention
  Acute haemodialysis patients
Daily values for creatinine, Unit: mg/dl or mmol/ or µmol/L | During the intervention
  Acute haemodialysis patients
Daily values for potassium, Unit: mg/dl or mmol/ or µmol/L | During the intervention
  Acute haemodialysis patients
Ultrafiltration volume (UF) and Effluent volume (per treatment) | During the intervention
  Acute haemodialysis patients
Values for urea and creatinine (measured according to the clinical practice of the site) | During the intervention
  Chronic haemodialysis patients
Planned and delivered UF-volume (per treatment) | During the intervention
  Chronic haemodialysis patients

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brauer, Dr. med., Principal Investigator — Jena University Hospital; Bernhard Schmidt, Prof Dr med, Principal Investigator — Hannover Medical School
Locations (2):
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena